CLINICAL TRIAL: NCT05241834
Title: A Phase 1 Study of Oral LOXO-260 in Patients With RET Fusion-Positive Solid Tumors, Medullary Thyroid Cancer, and Other Tumors With RET Activation Refractory to Selective RET Inhibitors
Brief Title: A Study of LOXO-260 in Cancer Patients With a Change in a Particular Gene (RET) That Has Not Responded to Treatment
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18381; J3T-OX-JZTA (Other: Eli Lilly and Company); LOXO-NGR-21001 (Other: Eli Lilly and Company)
Expanded Access: NCT05225259 (No longer available)
Record Dates: First submitted 2022-02-08; First posted 2022-02-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms
Keywords: Solid tumors with RET alteration
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1A: LOXO-260 Dose Escalation (Experimental): LOXO-260 administered orally
  Interventions: Drug: LOXO-260
- Phase 1B: LOXO-260 Dose Expansion (Experimental): LOXO-260 administered orally
  Interventions: Drug: LOXO-260

INTERVENTIONS:
Drug: LOXO-260 — Oral
  Other Names: LY3838915

SUMMARY:
The main purpose of this study is to learn more about the safety, side effects, and effectiveness of LOXO-260. LOXO-260 may be used to treat cancer that has a change in a particular gene (known as the RET gene). Participation could last up to 24 months (2 years) and possibly longer if the disease does not get worse.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years of age at the time of signing the informed consent (Phase 1a and Phase 1b). Patients 12 years and older may be enrolled in Phase 1b for countries and sites where approved.
* Must have evidence of a previously documented RET fusion (solid tumors) or RET mutation (MTC or MEN2-associated cancers) that is a histological or a cytological proven diagnosis of locally advanced, unresectable and/or metastatic cancer and meet cohort-specific criteria.
* Have received a prior selective RET inhibitor.
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 1 (age > 16 years), Karnofsky Performance Status (KPS) ≥ 80 (age > 16 years), or Lansky Performance Status (LPS) ≥ 40% (age < 16 years).
* Have discontinued all previous treatments for cancer with resolution of any significant AEs, and of all clinically significant toxic effects of prior locoregional therapy, surgery, radiotherapy, or systemic anticancer therapy.
* Have adequate organ function.
* Phase 1b expansion: Patients must have measurable disease per RECIST v 1.1.
* Phase 1b expansion: Molecular Pathology Results (including RET and other genes) from a sample, blood or tissue, taken on or after RET selective treatment.

Exclusion Criteria:

* Disease suitable for local therapy administered with curative intent.
* Have an active fungal, bacterial, and/or active untreated viral infection.
* The patient has a serious pre-existing medical condition(s).
* Have symptomatic CNS malignancy or metastasis.
* Patients treated with drugs known to be strong inhibitors or inducers of cytochrome P450 3A (CYP3A).
* Progression of disease within 4 months of starting a prior selective RET inhibitor.
* Phase 1b expansion: Patients harboring known activating bypass alterations outside RET that may confer resistance to LOXO-260.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1 a: To determine the MTD/RP2D of LOXO-260: Dose limiting toxicity (DLT) rate | During the first 28-day cycle of LOXO-260 treatment
  DLT rate

SECONDARY OUTCOMES:
Phase 1b: To assess the antitumor activity: Overall response rate (ORR) | Up to approximately 24 months or 2 years
  ORR per Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
To characterize the PK properties of LOXO-260: Mean concentration of LOXO-260 | Up to approximately 24 months or 2 years
  PK: Mean concentration of LOXO-260
To assess the antitumor activity of LOXO-260: ORR | Up to approximately 24 months or 2 years
  ORR per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Emin Avsar, Study Director — Eli Lilly and Company
Locations (16):
- United States (14):
  - UCLA Medical Center, Los Angeles, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Emory University, Atlanta, Georgia
  - University of Chicago Medicine-Comprehensive Cancer Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy (Igr), Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LOXO-260 in Cancer Patients with a Change in a Particular Gene (RET) that has not Responded to Treatment — https://trials.lillytrialguide.com/en-US/trial/4YkqlYP1cMtTbO3nqf7IKG